CLINICAL TRIAL: NCT00902200
Title: A Phase 2, Double-masked, Randomized, Placebo-controlled, Dose-response Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-12286 Ophthalmic Solution 0.05%, 0.1% and 0.25% in Patients With Elevated Intraocular Pressure
Brief Title: A Study of AR-12286 in Patient With Elevated Intraocular Pressure (IOP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-12286-CS201
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Elevated Intraocular Pressure
Keywords: Glaucoma; Intraocular pressure
MeSH Terms: conditions — Ocular Hypertension; Glaucoma | interventions — AR-12286

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vehicle (Placebo Comparator): q.d. (AM) x 7 days, then q.d. (PM) x 7 days, then b.i.d. x 7 days.
  Interventions: Drug: AR-12286 vehicle
- AR-12286 0.05% (Experimental): q.d. (AM) x 7 days, then q.d. (PM) x 7 days, then b.i.d. x 7 days.
  Interventions: Drug: AR-12286
- AR-12286 0.1% (Experimental): q.d. (AM) x 7 days, then q.d. (PM) x 7 days, then b.i.d. x 7 days.
  Interventions: Drug: AR-12286
- AR-12286 0.25% (Experimental): q.d. (AM) x 7 days, then q.d. (PM) x 7 days, then b.i.d. x 7 days.
  Interventions: Drug: AR-12286

INTERVENTIONS:
Drug: AR-12286 — See arms
  Arms: AR-12286 0.05%; AR-12286 0.1%; AR-12286 0.25%
Drug: AR-12286 vehicle — See arms
  Arms: Vehicle

SUMMARY:
Double-masked, randomized, multi-center, placebo-controlled parallel-comparison of AR-12286.

DETAILED DESCRIPTION:
Subjects will be randomized to receive AR-12286 Ophthalmic Solution 0.05%, 0.1%, and 0.25% or its vehicle (one eye), q.d. (AM) x 7 days, then q.d. (PM) x 7 days, then b.i.d. x 7 days. The first dose will be administered in the clinic. Ocular safety and ocular hypotensive efficacy will be evaluated in the clinic throughout this period.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater.
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT). Unmedicated (post-washout, if required) IOP >= 24 mm Hg in one or both eyes at 08:00 hours, >= 21 mm Hg at 10:00, 12:00 and 16:00 hours on post-washout measurement (Visit 1).
3. Corrected visual acuity in each eye +1.0 logMAR (logarithm mininum angle of resolution) or better by ETDRS (Early Treatment Diabetic Retinopathy Study) in each eye (equivalent to 20/200).
4. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

Either eye

1. Intraocular pressure > 36 mm Hg
2. Known hypersensitivity to any component of the formulation or to topical anesthetics, (benzalkonium chloride, etc.)
3. Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months.
4. History or evidence of ocular infection inflammation, or of herpes simplex keratitis, or clinically significant blepharitis or conjunctivitis at baseline (Visit 1)..
5. Contact lens wear within 30 minutes of instillation of study medication.
6. Ocular medication of any kind within 30 days of Visit 2, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after Visit 2) or c) lubricating drops for dry eye (which may be used throughout the study),
7. Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (i.e., cup-disc ratio > 0.8).
8. Central corneal thickness greater than 600 microns.
9. Any abnormality preventing reliable applanation tonometry.

   Study eye:
10. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure.

    Note: Previous laser peripheral iridotomy is acceptable.
11. Previous glaucoma intraocular surgery or laser procedures in study eye(s).
12. Refractive surgery in study eye(s) (e.g., radial keratotomy, PRK (photorefractive keratectomy), LASIK (Laser-Assisted in situ Keratomileusis), etc.).

    General/Systemic:
13. Clinically significant abnormalities in laboratory tests at screening (See Appendix 1).
14. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, cardiovascular or endocrine disorders) which might interfere with the study.
15. Participation in any investigational study within the past 30 days.
16. Changes of systemic medication during the study that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
17. Due to status of preclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be mean diurnal IOP on each day at which diurnal IOP is measured at each timepoint. | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tom van Haarlem, MD, Study Director — Aerie Pharmaceuticals, Inc.
Locations (8):
- United States (8):
  - Soilsh Practice, Pasadena, California
  - Bacharach practice, Petaluma, California
  - Hernando Eye Institute, Brooksville, Florida
  - Taustine Eye Center, Louisville, Kentucky
  - Mundorf Practice, Charlotte, North Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Texan Eye, Austin, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas

REFERENCES:
- [Derived] Williams RD, Novack GD, van Haarlem T, Kopczynski C; AR-12286 Phase 2A Study Group. Ocular hypotensive effect of the Rho kinase inhibitor AR-12286 in patients with glaucoma and ocular hypertension. Am J Ophthalmol. 2011 Nov;152(5):834-41.e1. doi: 10.1016/j.ajo.2011.04.012. Epub 2011 Jul 27. PMID 21794845